CLINICAL TRIAL: NCT05007431
Title: Violence Sexual Incidence During the First Year of Residence in the French Territory on Asylum Seekers in Marseille and Nice
Brief Title: Violence Sexual Incidence During the First Year of Residence on Asylum Seekers
Acronym: INCIDAVI
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-05
Record Dates: First submitted 2021-07-29; First posted 2021-08-16 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Sexual Violence
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women asylum seekers
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Data collection will be carried out by hetero-questionnaire carried out in the presence of the questioned.

SUMMARY:
Asylum seekers women are particularly exposed to sexual violence. One in seven women in France and one in three in the world say they have been a victim of sexual violence at least once in her life.

The main objective of this study is to measure the incidence of sexual violence suffered by women in asylum proceedings during their first year of stay on French territory, in Marseille and Nice.

DETAILED DESCRIPTION:
Introduction: One in seven women in France and one in three in the world say they have been a victim of sexual violence at least once in his life. They are exacerbated in vulnerable populations, marginalized, in post-conflict situations or population displacement.

Therefore asylum seekers women are particularly exposed to sexual violence. This is why OFPRA and the Ministry of Solidarity and Health have protected these women with regard to sexual violence, one of the priority issues for public health. Yet, the investigators do not know the proportion of women seeking asylum who have suffered violence on French soil. In addition, the investigators did not find an international study of the incidence of violence sexual abuse suffered in the host country by women seeking asylum. Objective: Determine the incidence of sexual violence that occurred in the year following the arrival on French soil of adult women in the asylum process in Marseille and Nice.

Methodology: Multicentric longitudinal observational study (Marseille and Nice) based on a historical cohort of sexual violence among women in the application process asylum. 1,800 adult women seeking asylum were registered in 2019 in Marseille and Nice. The number of subjects required is 450 women (1: 4 sample of the target population).

Data collection will be carried out by hetero-questionnaire carried out in the presence of the questioned.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years old
* Major arrival (> 18 years old) on French territory
* In the asylum application procedure with the GUDA in Marseille or Nice
* Having a decline of residence on French soil of twelve months over the last 2 years.
* No objection to participating in the study

Exclusion Criteria:

- Existence of cognitive disorders (dementia, mental retardation) limiting the collection of criteria for judgment

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women asylum seekers victims of sexual violence
Sampling Method: Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
Questionnaires on sexual violence suffered v1.1 | 6 months
  The incidence of any of the following four events: rape or attempted rape or sexual assault or sexual exhibition that occurred on French soil during the first year of residence in France with women in the asylum procedure in France, defined by at least one positive response on the questionnaire.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - AP-HM, Marseille
  - Chu de Nice, Nice

IPD SHARING:
Plan to Share IPD: No